CLINICAL TRIAL: NCT06524934
Title: The Impact of Virtual Reality Technology in the Era of See & Treat Hysteroscopy: A Randomized Controlled Trial
Brief Title: Virtual Reality's Role in See&Treat Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Brunella Zizolfi, Assistant Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 112/24
Record Dates: First submitted 2024-07-18; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Endometrial Cancer; Endometrial Diseases; Myoma;Uterus; Endometrial Hyperplasia
Keywords: Outpatient Hysteroscopy; Virtual Reality Technology; Pain and Anxiety Management; See & Treat
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Diseases; Myofibroma; Endometrial Hyperplasia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Experimental): The patients in this group undergo the procedure using virtual reality.
  Interventions: Device: Use of virtual reality during the hysteroscopic procedure
- Control group (No Intervention): The patients in this group undergo the procedure without the use of virtual reality.

INTERVENTIONS:
Device: Use of virtual reality during the hysteroscopic procedure — In VR group patients underwent hysteroscopy with standard care but the addition of VRT provided by a VR headset and headphones with the use of a Hypno VR software.
  Arms: Case group

SUMMARY:
The aim of the study is to evaluate the feasibility and effectiveness of virtual reality technology in outpatient hysteroscopy to improve pain and anxiety management and spread the diffusion of see & treat philosophy.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2024-07-06 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Pain pre procedure | 1 minute before the procedure
  Level of pain the patient thinks she will experience, expressed on a 10-point numerical rating scale (NRS), from 0 indicating no pain to 10 corresponding to the worst pain (subjective criteria), before undergoing diagnostic and operative procedures.
Anxiety pre procedure | 1 minute before the procedure
  Level of anxiety the patient thinks she will experience, expressed on a 10-point numerical rating scale (NRS), from 0 indicating no anxiety to 10 corresponding to the worst anxiety (subjective criteria), before undergoing diagnostic and operative procedures.
Pain post procedure | 1 minute after the procedure
  Level of pain reported by the patient, expressed on a 10-point numerical rating scale (NRS), from 0 indicating no pain or anxiety, to 10 corresponding to the worst pain (subjective criteria), during diagnostic and operative procedures.
Anxiety post procedure | 1 minute after the procedure
  Level of anxiety reported by the patient, expressed on a 10-point numerical rating scale (NRS), from 0 indicating no pain or anxiety, to 10 corresponding to the worst anxiety (subjective criteria), during diagnostic and operative procedures.
Heart rate (HR) pre procedure | 1 minute before the procedure
  Heart rate (HR) collected by a dedicate nurse before diagnostic or operative procedures (objective criteria).
Respiratory rate (RR) pre procedure | 1 minute before the procedure
  Respiratory rate (RR) collected by a dedicate nurse before diagnostic or operative procedures (objective criteria).
Heart rate (HR) during procedure | 5 minutes after the start of the procedure
  Heart rate (HR) collected by a dedicate nurse during diagnostic or operative procedures (objective criteria).
Respiratory rate (RR) during procedure | 5 minutes after the start of the procedure
  Respiratory rate (RR) collected by a dedicate nurse during diagnostic or operative procedures (objective criteria).

SECONDARY OUTCOMES:
Suspension rate of procedure | During procedure
  Procedure completion and suspension rate (defined as the proportion of suspended procedures for any reasons)
Time of procedure | During procedure
  Recording the time of procedure
Satisfaction rate | 5 minutes after the procedure
  Satisfaction rate (Virtual reality group: desire to use the headset again in the future / Control group: desire to use headset if they could)
Side effects | 5 minutes after the procedure
  Reported side effects

CONTACTS AND LOCATIONS:
Overall Officials: Brunella Ms Zizolfi, AssProfessor, Principal Investigator — University Federico II of Naples - Italy
Locations (1):
- University of Naples Federico II, Napoli, Italy